CLINICAL TRIAL: NCT04522791
Title: Breathing, Relaxation, Attention Training, & Health in Older Adults
Brief Title: Breathing, Relaxation, Attention Training, & Health in Older Adults (BREATHE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Stanford University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kathi Heffner, Associate Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00004727; R01NR015452 (NIH)
Record Dates: First submitted 2020-08-10; First posted 2020-08-21 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment; Healthy Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A double-blinded, phase II randomized controlled trial (RCT). Older adults with MCI (n=114) will be randomly assigned to an 8-week combined intervention (RFB+VSOP), VSOP with imagery-guided relaxation control (IR+VSOP), or a IR control (IR only), with 2-week booster sessions provided at 3- and 9-months after intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RFB+VSOP (MCI) (Experimental): For home-based RFB+VSOP: The investigators will instruct subjects to do 10-minutes of app- guided paced breathing at RF daily; for select days, there will be VSOP training immediately following RFB.
  A total of 8 weeks intervention. The investigators will extend the intervention for additional two weeks for make-up sessions.
  Interventions: Behavioral: RFB; Behavioral: VSOP
- IR+VSOP (MCI) (Active Comparator): The control IR strategy will be used, set-up of which will be the same as the RFB + VSOP intervention group with IR replacing RFB. A total of 8 weeks intervention. The investigators will extend the intervention for additional two weeks for make-up sessions.
  Interventions: Behavioral: VSOP; Behavioral: IR
- IR only (MCI) (Placebo Comparator): Participants randomized to this condition will receive weekly in-person check-in visits, and perform daily 10-minute IR, so that the number of treatment contacts (though not duration) will be equivalent. A total of 8 weeks intervention. The investigators will extend the intervention for additional two weeks for make-up sessions.
  Interventions: Behavioral: IR
- RFB+VSOP (HC) (Other): this is a new healthy control intervention arm used for testing adherence related items.
  For home-based RFB+VSOP: The investigators will instruct subjects to do 10-minutes of app- guided paced breathing at RF daily; for select days, there will be VSOP training immediately following RFB.
  A total of 8 weeks intervention. The investigators will extend the intervention for additional two weeks for make-up sessions.
  Interventions: Behavioral: RFB; Behavioral: VSOP

INTERVENTIONS:
Behavioral: RFB — The RFB protocol entails a combination of 8 weekly, in-lab training sessions using HRV biofeedback software (Physiocom, Seattle, WA) and daily paced breathing homework using a mobile-based HRV biofeedback app (Inner Balance, HeartMath, LLC, CA).
  Arms: RFB+VSOP (HC); RFB+VSOP (MCI)
Behavioral: VSOP — The investigators will use the INSIGHT online program (Posit Science). The platform will be built for our study, including 5 tasks (Eye for detail, Peripheral challenge, Visual sweep, Double decision, Target tracker) that practice different cognitive processes with PS/A as the shared domain.
  Arms: IR+VSOP (MCI); RFB+VSOP (HC); RFB+VSOP (MCI)
Behavioral: IR — Guided imagery relaxation, equal in dose and frequency to RF practice, will be used to control for relaxation effects that may occur via RFB (which could provide an alternative explanation for outcomes). IR activities will be facilitated using the Insight Timer mobile-based app, which emphasizes the use of visualization and imagery strategies to help the body relax.
  Arms: IR only (MCI); IR+VSOP (MCI)

SUMMARY:
A recently completed study suggested that processing speed and attention (PS/A) oriented cognitive training (VSOP) produced robust effect on PS/A and working memory, but not in cognitive control or episodic memory, and long-term effects were overall modest. The proposed R01 renewal proposes to identify additional attributes to further enhance transferred and long-term effects of PS/A training in older adults with amnestic mild cognitive impairment (MCI) by addressing adaptation capacity that underpins adaptive learning and neuroplasticity. The goal of the stage II double-blinded randomized trial is to test whether adding resonance frequency breathing (RFB) training to VSOP will strengthen multiple contributors to adaptation capacity, particularly the central and peripheral pathways of autonomic nervous system (ANS) flexibility, which will strengthen VSOP training effect on cognitive and brain function and slow the progress of dementia in MCI. The central hypothesis is that strengthening adaptation capacity, via improving autonomic nervous system (ANS) flexibility, will enhance neuroplasticity and slow progress of dementia in MCI, since adaptation capacity is critical for neuroplasticity of VSOP, but compromised in neurodegenerative process. Older adults with MCI (n = 114) will be randomly assigned to an 8-week combined intervention (RFB+VSOP), VSOP with guided imagery relaxation (IR) control, and a waitlist IR control, with periodical booster training sessions at follow-ups. Mechanistic and distal outcomes include ANS flexibility and multiple markers of dementia progress. Data will be collected across a 14-month period. The two primary aims are to examine long-term effects of the combined intervention on ANS flexibility (Aim 1), as well as the cognitive, behavioral, and functional capacity (Aim 2). The exploratory aim will be to determine the preliminary long-term effect of the combined intervention on neurodegeneration. This can be a reasonable renewal plan from the completed study, aiming to identify additional attributes to further enhance transferred and long-term effects of cognitive training in MCI. This will be among the first randomized controlled trials to examine a novel, combined intervention targeting adaptation capacity in MCI, with an ultimate goal for slowing neurodegeneration.

In addition, research on how to monitor adherence - the extent to which VSOP training is delivered and followed as intended - has been conceptually and methodologically limited. Robust monitoring of adherence to cognitive training requires valid assessment of effective engagement. Here, we apply our well-supported, novel framework of mental fatigability for measuring effective engagement in cognitive training. Mental fatigability, the failure to remain engaged in tasks requiring sustained mental effort, can be captured via measures of self-reported disengagement, increase in reaction time during tasks, and facial expression of negative valence/low arousal. These markers of disengagement relate to ventromedial prefrontal cortex dysfunction. We will apply this framework to advance understanding of the underpinnings of adherence to VSOP training by monitoring the extent of effective engagement while using the training platform.

ELIGIBILITY:
Inclusion Criteria:

1. All participants will require a diagnosis of "mild cognitive impairment due to Alzheimer's disease"using the most recent NIA and Alzheimer's Association workshop criteria:

   1. Presence of memory complaint,
   2. Rey Auditory Verbal Learning Test delayed recall (for memory) < 6,
   3. Montreal Cognitive Assessment (for global cognition) ranged 18 and 25,
   4. Activities of Daily Living Questionnaire ≤ 30,
2. Intact score for San Diego Brief Assessment of Capacity to Consent (UBACC).
3. If a participant is on Alzheimer's disease medication (i.e., memantine or cholinesterase inhibitors), antidepressants, anxiolytics, or vascular risk or diseases related medications (e.g., beta- blocker), the dose should be stable for 3 months prior to recruitment.
4. Age 60-89,
5. English-speaking,
6. Adequate visual and hearing acuity for using mobile-based apps and testing by self-report, and
7. Community-dwelling.

Exclusion Criteria:

1. Current enrollment in another cognitive improvement study;
2. Uncontrollable symptoms of major depression;
3. Major cerebrovascular and cardiovascular diseases (e.g., congestive heart failure, pacemaker, prior myocardial infarction);
4. Neurological diseases (e.g., Parkinson's disease, Multiple Sclerosis);
5. Having an active legal guardian (indicating impaired capacity for decision making);
6. MRI contraindication (e.g., pacemaker, claustrophobia).
7. Color blindedness
8. Alcohol dependency in the past 5 years that are the main contributor to MCI

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
change of ANS flexibility at 2 months from baseline | 2 months post-baseline
  A composite score developed via central autonomic networks and heart rate variability at rest and in response to a challenging cognitive stressor. Higher indicates better ANS flexibility. No max/min.
change of ANS flexibility at 8 months from baseline | 8 months post-baseline
  A composite score developed via central autonomic networks and heart rate variability at rest and in response to a challenging cognitive stressor. Higher indicates better ANS flexibility. No max/min.
change of ANS flexibility at 14 months from baseline | 14 months post-baseline
  A composite score developed via central autonomic networks and heart rate variability at rest and in response to a challenging cognitive stressor. Higher indicates better ANS flexibility. No max/min.
change of cognition at 2 months from baseline | 2 months post-baseline
  A composite score in executive function computed from Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER). No min/max; higher score indicates higher executive function. Z-transformation will be calculated.
  Visual episodic memory computed from Brief Visuospatial Memory Test-Revised (BVMT-R). Age normative percentile scores range from 0-100, higher indicating better memory. Z-transformation will be calculated.
  A composite score will be a mean Z-score of composite score of EXAMINER and percentile score of BVMT-R.
change of cognition at 8 months from baseline | 8 months post-baseline
  A composite score in executive function computed from Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER). No min/max; higher score indicates higher executive function. Z-transformation will be calculated.
  Visual episodic memory computed from Brief Visuospatial Memory Test-Revised (BVMT-R). Age normative percentile scores range from 0-100, higher indicating better memory. Z-transformation will be calculated.
  A composite score will be a mean Z-score of composite score of EXAMINER and percentile score of BVMT-R.
change of cognition at 14 months from baseline | 14 months post-baseline
  A composite score in executive function computed from Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER). No min/max; higher score indicates higher executive function. Z-transformation will be calculated.
  Visual episodic memory computed from Brief Visuospatial Memory Test-Revised (BVMT-R). Age normative percentile scores range from 0-100, higher indicating better memory. Z-transformation will be calculated.
  A composite score will be a mean Z-score of composite score of EXAMINER and percentile score of BVMT-R.

SECONDARY OUTCOMES:
change of instrumental activities of daily living function (IADL) at 2 months from baseline | 2 months post-baseline
  Timed IADL objectively measures performance speed and accuracy on multiple IADL domains. Time spent on each task will be recorded with adjustment on whether an individual accurately completed each task. Average completion time across the tasks will be used as the outcome measure; lower completion times indicate lower IADL function. No min/max
change of instrumental activities of daily living function (IADL) at 8 months from baseline | 8 months post-baseline
  Timed IADL objectively measures performance speed and accuracy on multiple IADL domains. Time spent on each task will be recorded with adjustment on whether an individual accurately completed each task. Average completion time across the tasks will be used as the outcome measure; lower completion times indicate lower IADL function. No min/max
change of instrumental activities of daily living function (IADL) at 14 months from baseline | 14 months post-baseline
  Timed IADL objectively measures performance speed and accuracy on multiple IADL domains. Time spent on each task will be recorded with adjustment on whether an individual accurately completed each task. Average completion time across the tasks will be used as the outcome measure; lower completion times indicate lower IADL function. No min/max

CONTACTS AND LOCATIONS:
Locations (1):
- Feng Lin, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin FV, Heffner K, Gevirtz R, Zhang Z, Tadin D, Porsteinsson A. Targeting autonomic flexibility to enhance cognitive training outcomes in older adults with mild cognitive impairment: study protocol for a randomized controlled trial. Trials. 2021 Aug 23;22(1):560. doi: 10.1186/s13063-021-05530-z. PMID 34425878